CLINICAL TRIAL: NCT02664493
Title: The Effect of Steroid Pulse Therapy for the Reduction of Acute Rejection Episode in Subclinical Borderline Changes: An Open-Label, Randomized Clinical Trial
Brief Title: The Effect of Steroid Pulse Therapy for the Reduction of Acute Rejection Episode in Subclinical Borderline Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Joo Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-10-017-002
Record Dates: First submitted 2016-01-14; First posted 2016-01-27 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Renal Failure
Keywords: kidney transplantation; subclinical borderline rejection; steroid pulse therapy
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SPT group (Experimental): The patients who will show borderline change in 2-week protocol biopsy with stable graft function will be included in this study.
  Methylprednisolone 0.5 g daily for 3 days will be administered in (Steroid pulse therapy) SPT group.
  Interventions: Drug: Methylprednisolone
- non-SPT group (No Intervention): The patients who will show borderline change in 2-week protocol biopsy with stable graft function will be included in this study.
  Steroid pulse therapy (SPT) will not be applied and no additional treatment will be added in non-SPT group

INTERVENTIONS:
Drug: Methylprednisolone — Steroid pulse therapy : Methylprednisolone 0.5 g daily for 3 days, followed by a tapered dose of 60 mg per day for a period of five days.
  Other Names: high dose steroid therapy
  Arms: SPT group

SUMMARY:
* Several studies have shown that about 30% of transplanted kidneys with stable function present with tubule-interstitial mononuclear cell infiltration in protocol biopsies and therefore meet criteria for acute rejection. This subclinical rejection (SCR) has also been correlated with subsequent chronic allograft nephropathy and allograft dysfunction.
* The Banff scheme defines the minimal threshold for acute T-cell mediated rejection as infiltration of 25% or more of the renal cortex with five or more mononuclear cells in a focus of tubulitis or intimal arteritis (histological indices i2t2 or v1) and refers to borderline changes as those with insufficient for a diagnosis of acute T-cell mediated rejection, including mild to moderate (<50%) cortical infiltration and one to four mononuclear cells per tubule in cross section (i1t1 or i2t1)
* No consensus for the treating patients with borderline changes has been reached. Borderline changes with graft dysfunction are occasionally routinely treated with steroid pulse and, whereas subclinical borderline changes are simply 'ignored'. Particularly, a previous study demonstrated that most cases designated borderline by histopathology are found to be non-rejection by molecular phenotyping
* The aim of this study is to investigate the effect of early steroid pulse therapy for the reduction of acute rejection episode during the first year after renal transplantation in the patients who will show subclinical borderline changes at 2-week protocol biopsy.

DETAILED DESCRIPTION:
Background

Several studies have shown that about 30% of transplanted kidneys with stable function present with tubule-interstitial mononuclear cell infiltration in protocol biopsies and therefore meet criteria for acute rejection (1). This subclinical rejection (SCR) has also been correlated with subsequent chronic allograft nephropathy and allograft dysfunction (2,3).

The Banff 97 working classification of renal allograft pathology was introduced to standardize the histological definition of acute allograft rejection and to guide treatment of renal transplant recipients (4,5). The Banff scheme defines the minimal threshold for acute T-cell mediated rejection as infiltration of 25% or more of the renal cortex with five or more mononuclear cells in a focus of tubulitis or intimal arteritis (histological indices i2t2 or v1) and refers to borderline changes as those with insufficient for a diagnosis of acute T-cell mediated rejection, including mild to moderate (<50%) cortical infiltration and one to four mononuclear cells per tubule in cross section (i1t1 or i2t1) (6).

The averaged prevalence of borderline SCR at 1-2 week is 24% (range 12-38%), at 1-2 months is 23% (range 21-27%), at 2-3 months is 23% (range 11-41%) and 1 year is 17% (range 7-44%) from selected studies (7). However, the pathogenic role of such limited cortical mononuclear infiltration is not well established and no consensus for the treating patients with borderline changes has been reached. In practice, borderline changes with graft dysfunction are occasionally routinely treated with steroid pulse and, whereas subclinical borderline changes are simply 'ignored'. Particularly, a previous study demonstrated that most cases designated borderline by histopathology are found to be non-rejection by molecular phenotyping (8). Furthermore, some previous studies have shown that the risk of infection is higher in patients receiving high dose steroid (9-12), and a previous study suggested that the infection risk was increased, up to as 1.5-fold, in patients receiving steroid pulse therapy (SPT) for acute rejection (13).

Some previous studies revealed that the graft survival rates with treated borderline SCR was 99.1% at 1-year, 95.1% at 5-years, and 93.7% at 10-years (14) and the graft survival rates with untreated borderline SCR was 90.9% at 1-year (15). However, there was no randomized controlled study on the effect of steroid pulse therapy in stable renal transplant recipients with subclinical borderline changes.

Purpose

* The reduction in risk of graft failure is the pivotal measure of effectiveness for evaluating immunosuppressive regimens for renal transplantation. However, because of the long follow-up periods and large sample size required for such an endpoint, randomized controlled trials of immunosuppressive therapies have mostly relied on the surrogate endpoints.
* In our institution, since routine protocol biopsies are performed at 2 weeks, 1 year, and 2 years after renal transplantation, it is practically difficult that graft survival is used as an endpoint for randomized controlled trials.
* From a meta-analysis for 31 observational studies (16), acute rejection was associated with an increased risk of graft loss risk ratios ranged from 1.2 - 10.5. Furthermore, chronic allograft nephropathy and graft survival is strongly correlated with acute rejection episode during the first year after renal transplantation (17,18).
* Therefore, the aim of this study is to investigate the effect of early steroid pulse therapy for the reduction of acute rejection episode during the first year after renal transplantation in the patients who will show subclinical borderline changes at 2-week protocol biopsy.
* To evaluate the benefit over the risk, this study also investigates the effect of early steroid pulse therapy on the opportunistic infection including bacterial, fungal, and viral infections.

ELIGIBILITY:
Inclusion Criteria:

The patients who fulfill all the following conditions

* Age 19 - 70 years.
* The patients who underwent renal transplantation.
* The patients who will show borderline change in 2-week protocol biopsy with stable graft function will be included in this study.

(Stable function is defined as serum creatinine ≤1.5 mg/dl and ≤15% increase in serum creatinine in the 2 weeks before biopsy.)

Exclusion Criteria:

* The patients who had clinical uremic symptom within 2 weeks after kidney transplantation..
* The patients who had elevated serum creatinine level more than 1.5mg/dl or 15% compared to previous result.
* The patients' age under 19 years or over 70 years.
* The patients who underwent preoperative desensitization.
* The patients who had multiple organ transplantation.
* The patients who showed an allergic reaction to steroid.
* The patients who had psychologic disease (eg. depression) or history of psychologic medication.
* The patients participated in another clinical trial within 30 days before this study.
* The patients who did not agree with a consent form.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The reduction of acute rejection episode during the first year after renal transplantation in the patients who will show subclinical borderline changes at 2-week protocol biopsy. | 1 year

SECONDARY OUTCOMES:
Persistent subclinical rejection and chronic graft nephropathy at 1 year protocol biopsy | 1 year
  the rejection will be defined according to Banff criteria including borderline rejection.
  the degree of chronic graft nephropathy will be calculated based on a chronic sum score of the sum of the Banff chronic indices (cg + ci + ct + cv).
  the persistent subclinical rejection rate and the degree of chronic graft nephropahty according to the groups will be compared.
The effect of early steroid pulse therapy on the opportunistic infection including bacterial, fungal, and viral infections. | 1 year
  infection episodes will be recorded.
  cytomegalovirus (CMV), BK polyomavirus (BKV), varicella zoster virus (VZV), bacteria, fungus, TB, pneumocystis carinii infection will be included.
  rate of infection according to groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Joo Kim, Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rush DN, Henry SF, Jeffery JR, Schroeder TJ, Gough J. Histological findings in early routine biopsies of stable renal allograft recipients. Transplantation. 1994 Jan;57(2):208-11. doi: 10.1097/00007890-199401001-00009. PMID 8310509
- [Result] Miyagi M, Ishikawa Y, Mizuiri S, Aikawa A, Ohara T, Hasegawa A. Significance of subclinical rejection in early renal allograft biopsies for chronic allograft dysfunction. Clin Transplant. 2005 Aug;19(4):456-65. doi: 10.1111/j.1399-0012.2005.00303.x. PMID 16008588
- [Result] Legendre C, Thervet E, Skhiri H, Mamzer-Bruneel MF, Cantarovich F, Noel LH, Kreis H. Histologic features of chronic allograft nephropathy revealed by protocol biopsies in kidney transplant recipients. Transplantation. 1998 Jun 15;65(11):1506-9. doi: 10.1097/00007890-199806150-00020. PMID 9645814
- [Result] Furness PN, Kirkpatrick U, Taub N, Davies DR, Solez K. A UK-wide trial of the Banff classification of renal transplant pathology in routine diagnostic practice. Nephrol Dial Transplant. 1997 May;12(5):995-100. doi: 10.1093/ndt/12.5.995. PMID 9175057
- [Result] Racusen LC, Solez K, Colvin RB, Bonsib SM, Castro MC, Cavallo T, Croker BP, Demetris AJ, Drachenberg CB, Fogo AB, Furness P, Gaber LW, Gibson IW, Glotz D, Goldberg JC, Grande J, Halloran PF, Hansen HE, Hartley B, Hayry PJ, Hill CM, Hoffman EO, Hunsicker LG, Lindblad AS, Yamaguchi Y, et al. The Banff 97 working classification of renal allograft pathology. Kidney Int. 1999 Feb;55(2):713-23. doi: 10.1046/j.1523-1755.1999.00299.x. PMID 9987096
- [Result] Solez K, Axelsen RA, Benediktsson H, Burdick JF, Cohen AH, Colvin RB, Croker BP, Droz D, Dunnill MS, Halloran PF, et al. International standardization of criteria for the histologic diagnosis of renal allograft rejection: the Banff working classification of kidney transplant pathology. Kidney Int. 1993 Aug;44(2):411-22. doi: 10.1038/ki.1993.259. PMID 8377384
- [Result] Nankivell BJ, Chapman JR. The significance of subclinical rejection and the value of protocol biopsies. Am J Transplant. 2006 Sep;6(9):2006-12. doi: 10.1111/j.1600-6143.2006.01436.x. Epub 2006 Jun 22. PMID 16796717
- [Result] de Freitas DG, Sellares J, Mengel M, Chang J, Hidalgo LG, Famulski KS, Sis B, Einecke G, Halloran PF. The nature of biopsies with "borderline rejection" and prospects for eliminating this category. Am J Transplant. 2012 Jan;12(1):191-201. doi: 10.1111/j.1600-6143.2011.03784.x. Epub 2011 Oct 12. PMID 21992503